CLINICAL TRIAL: NCT07370181
Title: Ketamine Irrigation Analgesia: For Controlling Postoperative Pain in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Ketamine Irrigation Analgesia in Laparoscopic Cholecystectomy
Acronym: Ketamine
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Makram Soliman, Associate Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04-2025-300750
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Pain
Keywords: ketamine; Postoperative pain; Laparoscopic Cholecystectomy
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Saline Solution; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group N (Placebo Comparator): Patients will receive the irrigation at the end of surgery after dissection; irrigation analgesia by 5 ml bupivacaine 0.50% plus 20 ml normal saline (Group N)
  Interventions: Drug: Normal saline
- Group K (Experimental): Patients will receive 5 ml bupivacaine 0.50% plus 1 mg/kg ketamine (Group K). The volume of irrigation in group K is completed by normal saline to reach a total of 25 ml.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Normal saline — Patients will receive the irrigation at the end of surgery after dissection; irrigation analgesia by 5 ml bupivacaine 0.50% plus 20 ml normal saline (Group N)
  Arms: Group N
Drug: Ketamine — Patients will receive 5 ml bupivacaine 0.50% plus 1 mg/kg ketamine (Group K). The volume of irrigation in group K is completed by normal saline to reach a total of 25 ml.
  Other Names: Katlar
  Arms: Group K

SUMMARY:
Patients will be assigned randomly to two groups (30 subjects each) to be anesthetized. The study drug will be delivered in opaque bags labeled "study drug" and 60 patients will be allocated in two groups (of 30 patients each) to receive the irrigation at the end of surgery after dissection; irrigation analgesia by 5 ml bupivacaine 0.50% plus 20 ml normal saline (Group N) or 5 ml bupivacaine 0.50% plus 1 mg/kg ketamine (Group K). The volume of irrigation in group K is completed by normal saline to reach a total of 25 ml.

DETAILED DESCRIPTION:
The anesthetic technique will be standardized for all groups. Anesthesia will be induced with propofol 2 mg.kg-1, fentanyl 1 µg.kg-1 and rocuronium 0.6 mg/kg1for muscle relaxation. The size of the cuffed endotracheal tube will be selected according to the patient's age. Anesthesia and muscle relaxation will be maintained with 2% sevoflurane in a 50% oxygen/air mixture and 0.1 mg/kg rocuronium at fixed intervals. All patients will receive volume-cycled mechanical ventilation in ventilator settings that maintained normocarbia. Intra-operatively, patients will receive IV paracetamol 15 mg/kg and 10 mL/kg infusions of normal saline. Hemodynamic data (HR and MBP) will be monitored during the intraoperative period but recorded at the end of surgery before drug irrigation (T0), after extubation (T1), at postoperative care unit PACU admission (T2), then 30 min (T3), 1 hour (T4) and 2 hours (T5). Blood glucose will be measured using a point-of-care device (ACCU-CHEK©, Roche Pharmaceuticals, Basel, Switzerland) before the start of irrigation (T0), at PACU admission (T1), then after 12 hours (T2) and 24 hours (T3) to assess the effect of study drugs on the stress response.

At the end of the procedure, the residual neuromuscular blockade will be reversed with standard doses of neostigmine and atropine. Patients will be extubated awake in the recovery position and transported to the Post Anesthesia Care Unit (PACU). The anesthesia time (time in minutes from induction of anesthesia till its discontinuation) and time to extubation (time in minutes from the discontinuation of anesthesia till extubation) will be recorded. After fulfilling the criteria for full recovery, patients will be transferred to the ward.

Postoperative pain was assessed at rest and at movement, using a 0-10 cm VAS pain scale, where 0=no pain and 10=the worst pain imaginable. According to the degree of pain given by the patient, the classification of severity was done as follows: No pain = 0, mild pain=1-3, moderate pain= 4-6, and severe pain ≥7. The pain was treated with a bolus of pethidine 1 mg/kg when the reported VAS pain scale is ≥ 4. The score was assessed at 0 (PACU admission), 1, 2, 4, 12, and 24 hours after surgery.

The time to first request rescue analgesia and the total consumption of postoperative rescue analgesics will be recorded. Any perioperative adverse events will be treated and recorded such as hypotension, bradycardia, desaturation (SpO2% < 92%), and postoperative vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age ≥18 years of ASA I-II who will be scheduled for elective laparoscopic cholecystectomy under general anesthesia.

Exclusion Criteria:

* History of congenital heart disease
* Hypertension
* Developmental delay, or
* Allergy to study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
The total consumption of rescue analgesics | 24 hours
  The total consumption of postoperative rescue analgesics was recorded from the time to first request rescue analgesia to patient discharge after 24 h.

SECONDARY OUTCOMES:
The VAS pain score | 24 hours
  Postoperative pain was assessed, using a 0-10 cm VAS pain scale, where 0=no pain and 10=the worst pain imaginable. According to the degree of pain given by the patient, the classification of severity was done as follows: No pain = 0, mild pain=1-3, moderate pain= 4-6, and severe pain ≥7.The pain was treated with a bolus of pethidine 1 mg/kg when the reported VAS pain scale is ≥ 4. The score was assessed at 0 (PACU admission), 1, 2, 4, 12, and 24 hours after surgery.
the time to first request for rescue analgesics | 24 hours
  The time to first request rescue analgesia will be recorded and treated with a bolus of pethidine 1 mg/kg when the reported VAS pain scale is ≥ 4 .

CONTACTS AND LOCATIONS:
Overall Officials: Omar Makram Soliman, MD, Study Director — Assiut University, Faculty of Medicine, Anesthesia, surgical ICU and pain management Department

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Saadati K, Razavi MR, Nazemi Salman D, Izadi S. Postoperative pain relief after laparoscopic cholecystectomy: intraperitoneal sodium bicarbonate versus normal saline. Gastroenterol Hepatol Bed Bench. 2016 Summer;9(3):189-96. PMID: 27458511; PMCID: PMC4947133.